CLINICAL TRIAL: NCT03467087
Title: Safety and Feasibility of Electrical Muscle Stimulation in Patients Undergoing Autologous and Allogeneic Stem Cell Transplantation or Chemotherapy Requiring Hospitalization
Brief Title: Safety and Feasibility of Electrical Muscle Stimulation During Stem Cell Transplantation or Intensive Chemotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Saarland (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: EMS-ICT-001
Record Dates: First submitted 2018-02-27; First posted 2018-03-15 (Actual); Last update posted 2018-03-15 (Actual); Status verified 2018-03

CONDITIONS: Electric Stimulation Therapy
Keywords: Stem cell transplantation; Chemotherapy; Rehabilitation; Electrical muscle stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (1):
- Electrical muscle stimulation (Experimental): Electrical muscle stimulation is administered on both thighs and upper arms using a Myopuls 2000D device. Pre-set training time is 30 minutes per day (15 minutes for thighs and 15 minutes for upper arms) for at least 5 days a week.
  Interventions: Device: Myopuls 2000D

INTERVENTIONS:
Device: Myopuls 2000D — Device: Myopuls 2000D (Curatec Services GmBH, 47443 Moers, Germany)

SUMMARY:
Intensive chemotherapy, with or without following autologous or allogeneic stem cell transplantation (HSCT), is often the only curative treatment option for patients with haematological malignancies, leave many survivors physically and psychologically impaired because of side effects, many caused by weeks of immobilisation. Electrical muscle stimulation (EMS) is a proven training tool to improve physical performance in seniors and patients with chronic disease. The investigators therefore intend to evaluate the safety and feasibility of EMS in patients undergoing autologous HSCT, allogeneic HSCT and intensive chemotherapy. To assess feasibility all patients are asked to document training time during hospitalization in an EMS diary.

Furthermore, physical Performance will be measured using the 6-minute-walking distance (6MWD) and Short Physical Performance Battery (SPPB) as well as psychological performance using the Multidimensional Fatigue Inventory (MFI) and EORTC QLQ-C30 at the start of chemotherapy (T1) and when patients are discharged from hospital (T2).

At the time intensive chemotherapy is started and all inclusion and no exclusion criteria are met, patients will receive an EMS device with electrodes and will be instructed on how to use the device. After that, baseline tests using the above mentioned tools will be performed.

EMS will be conducted with a "Myopuls 2000" (Curatec Services GmbH, Moers, Germany) device using 13 cm x 5 cm electrodes. Electrodes are placed subsequently on both thighs and upper arms with instructions to stimulate each limb for at least 15 minutes on at least 5 days per week. Stimulation settings were as follows: 300 µs pulse width, 60 Hz frequency, 5 seconds on, 5 seconds off. The amplitude is initially set to elicit a visible muscle contraction and patients are encouraged to increase the amplitude as much as tolerated. After an initial training session, patients are to use the devices on their own and document their activities in an EMS diary.

Patients are then asked to use EMS throughout their therapy in addition to physical therapy until the day of their discharge when the initially performed tests are repeated.

The investigators hypothesis is, that EMS can be safely applied in patients undergoing intensive chemotherapy regimens and that patients are able to administer EMS by themselfs.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 80 years of age
* ECOG mperformance status 0-2
* patients undergoing chemotherapy regimens and and expected hospitalization time of > 14 days

Exclusion Criteria:

* patients with pacemakers and defibrillators
* patients with metallic implants close to stimulation sites
* skin irritations and injuries at the site of electrode placement
* pregnancy
* epilepsy
* patient is physically or mentally unable to administer EMS by him/her -self
* history of ventricular arrhythmias
* peripheral arterial disease
* deep vein thrombosis in the past 3 month
* myocardial infarction or stroke in the past 3 month

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2016-02-03 (Actual); Primary Completion 2017-02-16 (Actual); Study Completion 2017-03-16 (Actual)

PRIMARY OUTCOMES:
Occurence of adverse events caused by EMS | through study completion, an average of 30 days
  Possible adverse events: bleeding events (defined according to the WHO Bleeding Scale ), arrhythmias, CK elevation, skin irritation
Feasibility of self administered EMS | At the time of discharge of every patients, after an average of 30 days
  Percentage of patients able to complete at least 2/3 of the pre-set training time

SECONDARY OUTCOMES:
Physical performance as assessed by the 6 minute walking distance | At the time of discharge of every patients, after an average of 30 days
  Patients were told to walk on a 40-meter floor with instructions to cover as much distance as possible in 6 minutes. Patients were allowed to stop and rest as often as necessary. Time was stopped by a technician who was also allowed to encourage participants with standardized phrases during the walk.
Physical performance as assessed by the Short Physical Performance Battery | At the time of discharge of every patients, after an average of 30 days
  The Short Physical Performance Battery as developed by Guralnik and colleagues ranges from 0 - 12 points with 0 points indicating the worst possible performance and 12 points as best result. The battery consists of 3 objective tests of lower body function with maximally 4 points to be reached in one test:
  1. A timed walk of 8 feet
  2. The time it takes to rise from a chair 5 times
  3. A standing balance test
Psychological performance as assessed by the Multidimensional Fatigue Inventory | At the time of discharge of every patients, after an average of 30 days
  The Multidimensional Fatigue Inventory (MFI-20) consists of 5 subscales including general, physical and mental fatigue, reduced motivation and reduced activity with 20 items in total (4 items per subscale). Each item is rated on a 5-point scale (1-5) and each subscale ranges from 4 to 20. Patients were asked to fill out the test form before or within 3 days from start of treatment (timepoint 1) and at the day of discharge (timepoint 2). Contrary to physical assessment, high scores in the MFI subscales mean greater fatigue and therefore worse psychological functioning.
Psychological performance as assessed by the EORTC QoL 30 questionnaire | At the time of discharge of every patients, after an average of 30 days
  The EORTC QOL-C30 questionnaire contains 30 items that are divided into five functional scales, three symptom scales, a global health status / Quality of Life (QoL) scale, and six single items. Functional scales assess physical function (ability to manage daily life), role function (at work and daily activities), emotional function (tension, anxiety, irritability and depression), social function (family life or social activities) and cognitive function (concentration and memory). Symptom scales ask for fatigue, nausea or pain and single items measure dyspnoea, insomnia, appetite loss, constipation, diarrhoea and financial impact. The global health status / QoL scale rates overall health and quality of life. Original data was processed according to the EORTC scoring manual into a 0- to 100-point scale. High scores in functional scales and QoL indicate adequate function and QoL. Patients with high scores on symptom scales and single items show more severe symptoms and impairments.

CONTACTS AND LOCATIONS:
Overall Officials: Moritz Bewarder, M.D., Principal Investigator — University Hospital, Saarland; Dominic Kaddu-Mulindwa, M.D., Principal Investigator — University Hospital, Saarland

IPD SHARING:
Plan to Share IPD: No
We do not plan to share individual participant data sets since we think there is no additional information to be gained from individual data sets in this very heterogenous group of patients

REFERENCES:
- [Background] Wiskemann J, Kleindienst N, Kuehl R, Dreger P, Schwerdtfeger R, Bohus M. Effects of physical exercise on survival after allogeneic stem cell transplantation. Int J Cancer. 2015 Dec 1;137(11):2749-56. doi: 10.1002/ijc.29633. Epub 2015 Jun 19. PMID 26061092
- [Background] Wiskemann J, Huber G. Physical exercise as adjuvant therapy for patients undergoing hematopoietic stem cell transplantation. Bone Marrow Transplant. 2008 Feb;41(4):321-9. doi: 10.1038/sj.bmt.1705917. Epub 2007 Nov 19. PMID 18026154
- [Background] Takekiyo T, Dozono K, Mitsuishi T, Murayama Y, Maeda A, Nakano N, Kubota A, Tokunaga M, Takeuchi S, Takatsuka Y, Utsunomiya A. Effect of exercise therapy on muscle mass and physical functioning in patients undergoing allogeneic hematopoietic stem cell transplantation. Support Care Cancer. 2015 Apr;23(4):985-92. doi: 10.1007/s00520-014-2425-7. Epub 2014 Sep 27. PMID 25256376
- [Background] Dobsak P, Novakova M, Fiser B, Siegelova J, Balcarkova P, Spinarova L, Vitovec J, Minami N, Nagasaka M, Kohzuki M, Yambe T, Imachi K, Nitta S, Eicher JC, Wolf JE. Electrical stimulation of skeletal muscles. An alternative to aerobic exercise training in patients with chronic heart failure? Int Heart J. 2006 May;47(3):441-53. doi: 10.1536/ihj.47.441. PMID 16823250
- [Background] Nuhr MJ, Pette D, Berger R, Quittan M, Crevenna R, Huelsman M, Wiesinger GF, Moser P, Fialka-Moser V, Pacher R. Beneficial effects of chronic low-frequency stimulation of thigh muscles in patients with advanced chronic heart failure. Eur Heart J. 2004 Jan;25(2):136-43. doi: 10.1016/j.ehj.2003.09.027. PMID 14720530
- [Background] Kern H, Barberi L, Lofler S, Sbardella S, Burggraf S, Fruhmann H, Carraro U, Mosole S, Sarabon N, Vogelauer M, Mayr W, Krenn M, Cvecka J, Romanello V, Pietrangelo L, Protasi F, Sandri M, Zampieri S, Musaro A. Electrical stimulation counteracts muscle decline in seniors. Front Aging Neurosci. 2014 Jul 24;6:189. doi: 10.3389/fnagi.2014.00189. eCollection 2014. PMID 25104935
- [Background] Windholz T, Swanson T, Vanderbyl BL, Jagoe RT. The feasibility and acceptability of neuromuscular electrical stimulation to improve exercise performance in patients with advanced cancer: a pilot study. BMC Palliat Care. 2014 May 1;13:23. doi: 10.1186/1472-684X-13-23. eCollection 2014. PMID 24808760
- [Derived] Bewarder M, Klostermann A, Ahlgrimm M, Bittenbring JT, Pfreundschuh M, Wagenpfeil S, Kaddu-Mulindwa D. Safety and feasibility of electrical muscle stimulation in patients undergoing autologous and allogeneic stem cell transplantation or intensive chemotherapy. Support Care Cancer. 2019 Mar;27(3):1013-1020. doi: 10.1007/s00520-018-4390-z. Epub 2018 Aug 9. PMID 30094730